CLINICAL TRIAL: NCT06461806
Title: Effect of Protein Source During Ketogenic Weight Loss Intervention on Lipid Metabolism and Inflammation
Brief Title: Effect of Protein Source During Ketogenic Weight Loss Intervention
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Concordia University, Montreal (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 90000185
Record Dates: First submitted 2024-05-30; First posted 2024-06-17 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Obesity; Obesity; Endocrine
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: Participant are randomized to a plant or animal protein based ketogenic diet for a 12 week period. They are provided with the plant or animal proteins which they consume in the form of a smoothie twice a day. The remaining meal comprises of self selected foods.
Who Masked: Participant
Masking Description: Participants are provided with unlabelled protein containers in this single-blind study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plant-based pea/lupine protein supplement (Experimental)
  Interventions: Dietary Supplement: Protein supplement - Plant protein
- Animal-based whey protein supplement (Experimental)
  Interventions: Dietary Supplement: Protein supplement - Animal protein

INTERVENTIONS:
Dietary Supplement: Protein supplement - Plant protein — Pea/lupine protein powder mix
  Arms: Plant-based pea/lupine protein supplement
Dietary Supplement: Protein supplement - Animal protein — Whey protein powder
  Arms: Animal-based whey protein supplement

SUMMARY:
This randomized, controlled, single-blinded study will investigate how the protein source in a high-protein ketogenic diet affects metabolic weight loss outcomes after a 12-week dietary intervention

DETAILED DESCRIPTION:
This randomized, controlled, single-blinded study will compare how a ketogenic weight loss diet, supplemented with either animal- or plant-based protein affects: (i) metabolic markers (adipokine and cytokine) in adipose tissue and blood, (ii) adipose tissue immune cell profiles, and (iii) adipocyte characteristics and their interaction with other cells (e.g. immune cells and muscle cells). To better determine how tissue characteristics affect the whole body level, the relationships between adipose tissue characteristics and blood lipid and inflammatory markers will also be examined. Participants undergo anthropometric measurements, questionnaires, body composition assessment, energy assessment, blood draws, and adipose tissue biopsies from the abdominal and femoral adipose tissue depots

ELIGIBILITY:
Inclusion Criteria:

* Adults between 18-60 years old
* BMI: >29.99kg/m2

Exclusion Criteria:

* Any chronic metabolic conditions (e.g. CVD)
* Renal impairment (creatinine clearance <60 mL/min)
* Uncontrolled hypothyroidism
* Pregnant, breastfeeding, or postmenopausal females
* Past (<6 year) or present use of nicotine products
* Use of cannabis products
* Use of any other medications that may affect study outcomes (e.g. anti-depressants)
* Participants who have had a number of CT scans in the course of the year
* Participants following a vegan diet

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Change in weight | Baseline and at 12 weeks
  Overall weight loss, kg
Change in BMI | Baseline and at 12 weeks
  Height and weight will be combined to report BMI (kg/m^2)
Change in fat mass | Baseline and at 12 weeks
  Body composition is measured by dual energy x-ray absorptiometry.
Change in overall body fat percentage | Baseline and at 12 weeks
  Body composition is measured by dual energy x-ray absorptiometry.
Regional subcutaneous adipose tissue immune cells ( number of cells per gram tissue, percentage of the stromal vascular compartment) | Baseline and at 12 weeks
  Changes in various adipose tissue immune cells including M1-like and M2-like macrophages, T helper cells, and cytotoxic T cells will be measured via flow cytometry.
Concentrations of Circulatory cytokines and adipokines | Baseline and at 12 weeks
  Changes in cytokines and adipokines will be measured via ELISA. We will measure markers including interleukin 6, tumour necrosis factor a, leptin, and adiponectin.
Resting energy expenditure | Baseline and at 12 weeks
  Resting energy expenditure will be measured in a fasted state by indirect calorimetry. Volume of oxygen and carbon dioxide and water vapor pressure will be taken into consideration to calculate the resting energy expenditure.
Substrate oxidation | Baseline and at 12 weeks
  Substrate oxidation will be measured in a fasted state by indirect calorimetry. Volume of oxygen and carbon dioxide and water vapor pressure will be taken into consideration to calculate the respiratory exchange ratio.
Lipidomics | Baseline and at 12 weeks
  Lipidomics will be measured by mass spectrometry.
Adipocyte size | Baseline and at 12 weeks
  Regional adipocyte characteristics will be measured in vitro including adipocyte size,
Rate of pre-adipocyte proliferation | Baseline and at 12 weeks
  Regional adipose tissue pre-adipocyte proliferation rate will be measured in vitro

CONTACTS AND LOCATIONS:
Overall Officials: Sylvia Santsa, PhD, Principal Investigator — Concordia University, Montreal
Locations (1):
- School of Health, Concordia University, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
On request and approval by ethics
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data will be available after the study results have been accepted for publication. The data will be available for 5 y.
Access Criteria: On request with ethics approval.